CLINICAL TRIAL: NCT00637793
Title: A Double-Blind, Placebo-Controlled, Cross Over Study Using a Latin Square Design to Evaluate the Safety, Tolerability, and Efficacy of NGX267 Oral Capsules in Patients With Xerostomia Associated With Sjogren's Syndrome
Brief Title: Study of NGX267 Oral Capsules in Patients With Xerostomia Associated With Sjorgren's Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: TorreyPines Therapeutics (Industry)
Responsible Party: Susan Mellberg, R.N., M.B.A.; VP, Project Management, TorreyPines Therapeutics, Inc.
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: NGX267XSS2001
Record Dates: First submitted 2008-03-11; First posted 2008-03-18 (Estimated); Last update posted 2009-01-29 (Estimated); Status verified 2009-01

CONDITIONS: Xerostomia; Sjogren's Syndrome
Keywords: Xerostomia; Sjogren's Syndrome
MeSH Terms: conditions — Xerostomia; Sjogren's Syndrome | interventions — (S)-2-ethyl-8-methyl-1-thia-4,8-diazaspiro(4.5)decan-3-one

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Placebo Comparator): Placebo capsules
  Interventions: Drug: NGX267
- 2 (Experimental): 2 capsules in the am of each treatment period
  Interventions: Drug: NGX267
- 3 (Experimental): 2 capsules in the am of each treatment period
  Interventions: Drug: NGX267
- 4 (Experimental): 2 capsules in am of each treatment period
  Interventions: Drug: NGX267

INTERVENTIONS:
Drug: NGX267 — 2 capsules in the am of each treatment period
  Arms: 2
Drug: NGX267 — 2 capsules in the am of each treatment period
  Arms: 3
Drug: NGX267 — 2 capsules in the am of each treatment period
  Arms: 1
Drug: NGX267 — 2 capsules in the am of each treatment period
  Arms: 4

SUMMARY:
The purpose of this study is to evaluate the effectiveness of NGX267 in the improvement of decreased salivary flow associated with primary or secondary Sjögren's syndrome.

For each patient, the study includes four periods of treatment separated by a washout period that may range from 4 - 8 days according to patient and site discretion. Each treatment period includes two overnight stays in the clinic. One dose of study drug is taken during each treatment period

ELIGIBILITY:
Inclusion Criteria:

* Males and females aged 21 to 55 years, diagnosed with primary or secondary Sjögren's syndrome.
* Patients with a complaint of dry mouth based upon difficulty in speaking, swallowing, a sensation of mouth or throat dryness, lip or tongue dryness, or a level of thirst of sufficient intensity for the patient to seek therapy.
* Females of childbearing potential must not be at risk for pregnancy during the study. Females not of childbearing potential include postmenopausal and women who have been surgically sterilized.
* Patients must not be in an acute phase of illness.

Exclusion Criteria:

* Patients who have clinically significant reduction kidney function. cardiovascular abnormalities; lymphoma secondary to Sjögren's syndrome; pulmonary disease; the presence of enlarged salivary glands; physical closure of the salivary gland or known surgical procedure on the lacrimal punctum.
* Patients with diagnoses of a current gastrointestinal (GI) disease that would be exacerbated by the use of cholinomimetics; a current and acute psychiatric disorder, acute iritis, narrow angle glaucoma, or retinal disease as determined by medical history and physical examination.
* Patients who are otherwise judged inappropriate for inclusion in the study by the investigator
* Patients who have received any experimental drugs or devices or participated in any clinical trial within 30 days prior to screening including participation in a previous NGX267 clinical trial.
* Patients who are allergic to compounds that are similar to NGX267.

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2008-02; Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Quantitative and qualitative assessment of dry mouth | 36 days

SECONDARY OUTCOMES:
Tolerability and safety of NGX267 | 36 days

CONTACTS AND LOCATIONS:
Overall Officials: Walter F. Chase, M.D., Principal Investigator — Walter F. Chase MD. PA; Alan Kivitz, M.D., Principal Investigator — Altoona Center for Clinical Research; Frederick B. Vivino, M.D., Principal Investigator — Penn Rheumatology Associates and Sjogren's Syndrome Center
Locations (3):
- United States (3):
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania
  - Penn Rheumatology Associates and Sjogren's Syndrome Center, Philadelphia, Pennsylvania
  - Walter F. Chase MD PA, Austin, Texas